CLINICAL TRIAL: NCT04834765
Title: Using the Arts as a Proactive Mental Health Strategy for Generation Z
Brief Title: Mindfulness-Based Art Therapy and Generation Z
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Theresa Van Lith, Associate Professor & Clinical Coordinator of Art Therapy, Florida State University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: TVanLith
Record Dates: First submitted 2021-03-17; First posted 2021-04-08 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Anxiety Depression
Keywords: Stress

STUDY DESIGN:
Intervention Model Description: 3 intervention groups- Mindfulness only, Art Therapy only and combined Mindfulness based Art Therapy. 1 control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mindfulness (Active Comparator): Participants will be engaging in a mindfulness tasks twice per week for 5 weeks in which they will learn techniques through the use of yoga, meditation and breathwork.
  Interventions: Other: Mindfulness-only
- Art Therapy (Active Comparator): Participants will engage in art therapy with the use of clay twice per week through prompts.
  Interventions: Other: Art-only
- Mindfulness based Art Therapy (Active Comparator): Participants will engage in both mindfulness activities and art therapy twice per week and will learn techniques through the use of yoga, mediation, breathwork and art.
  Interventions: Other: Mindfulness-based art therapy
- Control Group (No Intervention): Participants will go about daily life as usual.

INTERVENTIONS:
Other: Mindfulness-based art therapy — The researchers developed a novel MBAT intervention consisting of 10 easily reproducible, clay-based MBAT directives, administered through an online platform delivery strategy. By developing an MBAT intervention that uses an online delivery strategy, the researchers realized it may have the potential of decreasing demands placed on counseling centers.
  Arms: Mindfulness based Art Therapy
Other: Art-only — The AO modules consist of an open-ended art-making exercise, with minimal direction. The AO intervention is designed as an 'art for art's sake' intervention with the focus on the art-making and less on outcome or product. Participants are asked to pull their ball of clay out and spend ten minutes creating a form from the clay to visually express their experience in the present moment.
  Arms: Art Therapy
Other: Mindfulness-only — The MO modules consist of only the mindfulness practices from the ABM intervention. The participants to follow along with a five-minute light yoga sequence, where asanas (yoga postures) are cued with breath. Yoga, for the purposes of the study, is explicitly defined to participants as the unity of breath with body movement. Poses were chosen based on their accessibility to a variety of body types and abilities, and chosen because they are documented to aid in grounding, increased haptic awareness, lowered levels of stress and anxiety, and restoration.
  Arms: Mindfulness

SUMMARY:
A randomized controlled trial will be conducted to determine the unique role of the arts as a proactive mental health strategy for college students in Generation Z. Arts-only, mindfulness-only, and arts-based mindfulness interventions as they compare to a non-intervention control group. These interventions will be delivered using a minimal contact, web-based approach. Psychological and physiological outcomes will be measured to determine if arts-related interventions activate unique and distinguishable mechanisms of change compared to the mindfulness only intervention and non-intervention control groups. In addition, protective effects will be assessed based on student participants' response to an acute academic stress simulation. Qualitative data in the form of transcribed exit interviews will be analyzed to characterize the unique needs of Generation Z students, along with level of engagement, intervention acceptance and satisfaction.

DETAILED DESCRIPTION:
To reach the general population of college students, a technology-assisted approach is paramount. This multidisciplinary project will tease apart the mechanisms of change and implications of employing art therapy approaches for anxiety and stress reduction in college students at much more nuanced level than previously tested using the MBAT approach designed and comparing it to its main components as isolated interventions.

Based on the previous two studies and the accumulated research explored, the following study aims and hypotheses will guide the proposed study.

These are:

Aim 1. To examine the psychological and physiological differences between an Mindfulness-based Art Therapy (MBAT) intervention, its components as isolated Art-Only (AO) and Mindfulness-Only (MO) interventions, and a non-intervention control (C) using a minimal contact, web-based approach with students in Generation Z. Hypothesis 1: MBAT, AO, and MO will produce distinguishable differences in participant outcomes related to anxiety and stress symptomology, protective factors against chronic stress, and the biological stress response compared to a non-intervention control. Aim 2. To evaluate how these interventions affect participants' responses to an acute academic stress simulation using the TSST paradigm. Hypothesis 2: Results of self-report assessments and saliva samples collected during the acute academic stress simulation will produce distinguishable differences between group conditions, suggesting that the art-based interventions engage unique mechanisms of change compared to the Mindfulness-Only intervention. Aim 3. To determine which intervention produces the greatest participant satisfaction and acceptance. Hypothesis 3: Participants of the MBAT and AO interventions will report higher levels of study engagement, overall study satisfaction, and intervention acceptance compared to participants of the MO intervention and non-intervention control group conditions.

B. Research Design The study will investigate the fundamental science underlying MBAT, a specific evidence-based form of therapy that includes mindfulness practices like meditation and yoga, and art therapy. The application of MBAT as a proactive mental health strategy in a pragmatic real-world setting is urgently needed, particularly given the stigma that surrounds mental health. The multidisciplinary team includes detailed expertise in art therapy, clinical psychology, mindfulness, and biological mechanisms. The study will involving using simple but validated psychological and biological measures to evaluate relatively brief, technology-assisted art-based mindfulness.

The study will involve conducting a randomized control research design to meet the specific aims proposed. College students will be randomized into one of four group conditions: 1) MBAT; 2) AO; 3) MO; or 4) C. Interventions will be administered using Canvas, the pre-existing learning management system of Florida State University. Students will be able to join the study on Canvas, complete the self-report measures, and receive nearly all of the intervention material virtually, eliminating several of the issues with current mental health programs.

There are no studies that specifically examine the effects of mindfulness based art therapy on inflammation or stress mediators besides our preliminary findings (Beerse et al., 2019). Biological research in art therapy to date has been limited to cortisol analysis alone, with a focus on the impact of different art materials on physiological stress. The proposed study will identify several interrelated biological systems influenced by the intervention and position us to isolate key mechanistic processes. Importantly, the study will involve using non-invasive biological sampling of saliva and will use the TSST to mimic acute academic stress; neither approach has been applied to MBAT. Additionally, minimal research has been conducted on the application of MBAT with young adults except studies related to serious health diagnoses such as cancer, palliative care, or heart disease. Therefore, this project addresses this gap in research using a research strategy that studies a general population, ensures easy reproducibility, and promotes the advancement of related innovative practices in arts research. The proposed approach thus has the potential to innovate the delivery of a cost-effective and efficacious alternative therapy that could reduce the societal burden of mental health symptoms and build resiliency among young adults.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled full time in an academic program at Florida State University and fit within age category of Generation Z

Exclusion Criteria:

* Regular tobacco smoking and over the age of 25

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2020-04-05 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-04-05 (Actual)

PRIMARY OUTCOMES:
IL-6 Saliva Elisa | Change from Week 1 to twice during Week 5 conducted before and after TSST
  Tests for levels human Interleukin-6
Salimetrics Cortisol EIA Test | Change from Week 1 to twice during Week 5 conducted before and after TSST
  Tests for salivary cortisol levels

SECONDARY OUTCOMES:
Generalized Anxiety Disorder 7 (GAD-7)- Spitzer et al. 2006 | Within first four weeks before study commences, then change from Week 1, to during Week 5, and then to 6 week follow-up
  Assesses anxiety symptoms. Each item is scored on a four-point Likert scale (0-3) with total scores ranging from 0 to 21 with higher scores reflecting greater anxiety severity. Scores above 10 are considered to be in the clinical range.
Somatic Symptom Scale 8 (SSS-8)- Gierk et al. 2014 (A brief version of the popular Patient Health Questionnaire - 15) | Change from Week 1, to during Week 5, and then to 6 week follow-up
  Assesses presence and severity of common somatic symptoms. A score of 0 to 3 points were classified as "no to minimal" severity, a score of 4 to 7 points as "low," a score of 8 to 11 points as "medium," a score of 12 to 15 points as "high," and a score of 16 points or higher as "very high."
Pittsburgh Sleep Quality Index (PSQI)- Buysse 1989 | Change from Week 1, to during Week 5, and then to 6 week follow-up
  Assesses sleep quality. The PSQI includes a scoring key for calculating a patient's seven sub scores, each of which can range from 0 to 3. The sub scores are tallied, yielding a "global" score that can range from 0 to 21. A global score of 5 or more indicates poor sleep quality; the higher the score, the worse the quality.
5 Facet Mindfulness Questionnaire Short Form (FFMQ)- Bohlmeijer et al. 2011 | Change from Week 1, to during Week 5, and then to 6 week follow-up
  Assesses 5 facets of mindfulness- observation, description, awareness of actions, non-judgement and non-reaction. Items scored on a 5-point Likert-type scale ranging from 1 (never or very rarely true) to 5 (very often or always true). Facet scores were computed by summing the scores on the individual items. Facet scores range from 8 to 40 (except for the nonreactivity facet, which ranges from 7 to 35), with higher scores indicating more mindfulness.
Perceived Stress Scale 10 (PSS-10)- Cohen, Kamarck and Mermelstein 2016 | Change from Week 1, to during Week 5, and then to 6 week follow-up
  Assesses perceptions of stress. PSS-10 scores are obtained by reversing the scores on the four positive items, e.g., 0=4, 1=3, 2=2, etc. and then summing across all 10 items. Items 4,5, 7, and 8 are the positively stated items.
Patient Health Questionnaire 9 (PHQ-9)- Kroenke et al. 1999 | Change from Week 1, to during Week 5, and then to 6 week follow-up
  Measures depression severity. This is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 0- not at all, 1- several days, 2- more than half the days, 3- nearly every day, respectively. PHQ-9 total score for the nine items ranges from 0 to 27. 1-4 minimal depression, 5-9 mild depression, 10-14 moderate depression, 15-19 moderately severe depression, 20-27 severe depression.
Oldenburg Burnout Inventory (OBI)- Demerouti & Bakker 2007 | Change from Week 1, to during Week 5, and then to 6 week follow-up
  Assesses burnout via disengagement and exhaustion. The subject is presented with a series of 16 statements, which they may agree or disagree with and is asked to indicate the degree of agreement or disagreement. The 16 items are divided between two subscales, the items are also summed to form two sub-totals. Disengagement items: 1, 3, 6, 7, 9, 11, 13 and 15; Exhaustion items: 2, 4, 5, 8, 10, 12, 14 and 16. For items 2, 3, 4, 6, 8, 9, 11 and 12, the scale is reversed, with Strongly Agree answers scoring 4 and Strongly Disagree answers scoring 1.
  A total OLBI score can be reached by summing the two sub-totals. The higher the score, the greater the level of burnout. Some therapists may categorize the OLBI scores under low, medium or high but no widespread consensus exists.
The DSM-5 Level 1 Cross-Cutting Symptom Measure (DSM5_Level 1) | Within first four weeks before study commences
  Consists of 23 questions that assess 13 psychiatric domains, including depression, anger, mania, anxiety, somatic symptoms, suicidal ideation, psychosis, sleep problems, memory, repetitive thoughts and behaviors, dissociation, personality functioning, and substance use. Nineteen of the 25 items on the measure are each rated on a 5-point scale (0=none or not at all; 1=slight or rare, less than a day or two; 2=mild or several days; 3=moderate or more than half the days; and 4=severe or nearly every day). The higher the score the more severity of the symptoms. The suicidal ideation, suicide attempt, and substance abuse items are each rated on a "Yes, No, or Don't Know" scale.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Van Lith, PhD, Principal Investigator — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States

REFERENCES:
- [Derived] Van Lith T, Cheshure A, Pickett SM, Stanwood GD, Beerse M. Mindfulness based art therapy study protocol to determine efficacy in reducing college stress and anxiety. BMC Psychol. 2021 Sep 3;9(1):134. doi: 10.1186/s40359-021-00634-2. PMID 34479649

DOCUMENTS (1):
  • Informed Consent Form (2020-08-31): https://cdn.clinicaltrials.gov/large-docs/65/NCT04834765/ICF_000.pdf